CLINICAL TRIAL: NCT00856141
Title: In Vivo Evaluation of Dynamic IOP Measuring Device During Phacoemulsifcation: A Prospective Randomised Clinical Trial
Brief Title: Set up for in-Vivo Measurement of Dynamic Intraocular Pressure (IOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: DR. SHETAL RAJ, ICIRC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 005-036; IOP set up; IOP fluctuations
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Intraocular Pressure
Keywords: IOP measurement; IOP fluctuation; in-vivo IOP measuring device; intraocular pressure measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. High fluidic parameters (Experimental): Bottle height varied from 90-110cms, fixed aspiration flow rate 40cc/min, vacuum upto 650mmHg depending on the grade of cataract
  Interventions: Device: phacoemulsifcation
- 2. Low fluidic parameters (Active Comparator): Bottle height varied from 70-90cms, fixed aspiration flow rate of 25cc/min, vacuum upto 400mmHg, depending on the grade of cataract
  Interventions: Device: phacoemulsifcation

INTERVENTIONS:
Device: phacoemulsifcation — A sensor (Blumenthal cannula) connected to a transducer, a signal amplifier, an IOP recording device, and a display unit
  Other Names: high aspiration flow rate,; high vacuum
  Arms: 1. High fluidic parameters
Device: phacoemulsifcation — A sensor (Blumenthal cannula) connected to a transducer, a signal amplifier, an IOP recording device, and a display unit
  Other Names: low flow rate; low vacuum; low bottle height
  Arms: 2. Low fluidic parameters

SUMMARY:
In this modern era, surgeons prefer to perform emulsification through small micro incisions. To accomplish this safely, surgeons raise irrigation bottle heights or use forced infusion systems.We believe that this sustained rise in the IOP during micro-incision phacoemulsification for a substantial period could be detrimental to the ocular structures. Therefore, intra-operative IOP pertaining to micro-incision cataract surgery is an emerging concern.

Conventional systems for measuring IOP generate an isolated graph of continuous pressure recording. Interpretation of the IOP fluctuations from these graphs requires a two step superimposition approach to characterize the IOP changes.

DETAILED DESCRIPTION:
The aim of the present study was to describe a new setup for intra-operative monitoring of IOP in a clinical setting and validate it by correlating IOP differences arising with different phacoemulsification parameters in eyes undergoing microincision coaxial phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing phacoemulsification for uncomplicated senile cataracts
* Cataracts from grade 1 to 3

Exclusion Criteria:

* presence of glaucoma,
* diabetic retinopathy,
* retinal vascular disease,
* high myopia (defined as AL > 25mm),
* uveitis,
* previous ocular trauma or surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
IOP fluctuation during each phase of surgery | intra-operative

SECONDARY OUTCOMES:
comparison of IOP fluctuations between high and low parameters group | intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Abhay R Vasavada, FRCS, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- Raghudeep Eye Clinic, Ahmedabad, Gujarat, India

REFERENCES:
- [Background] Grinbaum A, Blumenthal M, Assia E. Comparison of intraocular pressure profiles during cataract surgery by phacoemulsification and extracapsular cataract extraction. Ophthalmic Surg Lasers Imaging. 2003 May-Jun;34(3):182-6. PMID 12757089
- [Background] Georgescu D, Payne M, Olson RJ. Objective measurement of postocclusion surge during phacoemulsification in human eye-bank eyes. Am J Ophthalmol. 2007 Mar;143(3):437-40. doi: 10.1016/j.ajo.2006.11.017. Epub 2006 Dec 18. PMID 17222793
- [Background] Khng C, Packer M, Fine IH, Hoffman RS, Moreira FB. Intraocular pressure during phacoemulsification. J Cataract Refract Surg. 2006 Feb;32(2):301-8. doi: 10.1016/j.jcrs.2005.08.062. PMID 16565009
- [Background] Moorhead LC, Gardner TW, Lambert HM, O'Malley RE, Willis AW, Meharg LS, Moorhead WD. Dynamic intraocular pressure measurements during vitrectomy. Arch Ophthalmol. 2005 Nov;123(11):1514-23. doi: 10.1001/archopht.123.11.1514. PMID 16286613
- [Background] Joos KM, Kay MD, Pillunat LE, Harris A, Gendron EK, Feuer WJ, Steinwand BE. Effect of acute intraocular pressure changes on short posterior ciliary artery haemodynamics. Br J Ophthalmol. 1999 Jan;83(1):33-8. doi: 10.1136/bjo.83.1.33. PMID 10209431